CLINICAL TRIAL: NCT01627561
Title: Safety and Immunogenicity of GSK Biologicals' HPV-16/18 L1 VLP AS04 Vaccine (GSK-580299) in Healthy Female Children 4-6 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 115887; 2011-005604-15 (EudraCT Number)
Record Dates: First submitted 2012-06-14; First posted 2012-06-26 (Estimated); Results first posted 2015-05-08 (Estimated); Last update posted 2020-04-10 (Actual); Status verified 2020-03

CONDITIONS: Infections, Papillomavirus
Keywords: Immune response; Human papillomavirus; HPV vaccine; Safety
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18; Measles-Mumps-Rubella Vaccine; Diphtheria-Tetanus-acellular Pertussis Vaccines; Pentetic Acid

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Cervarix Group (Experimental): Healthy female subjects aged between, and including, 4 and 6 years, who received two doses of Cervarix vaccine at Day 0 and Month 6, administered intramuscularly in the deltoid muscle of the left upper arm.
  Interventions: Biological: Cervarix
- Priorix + Infanrix Group (Active Comparator): Healthy female subjects aged between, and including, 4 and 6 years, who received one dose of Priorix vaccine at Day 0 and one dose of Infanrix vaccine at Month 6, administered intramuscularly in the deltoid muscle of the left upper arm.
  Interventions: Biological: Priorix; Biological: Infanrix

INTERVENTIONS:
Biological: Cervarix — 2 doses administered intramuscularly in the deltoid muscle of the left arm at Day 0 and Month 6.
  Other Names: HPV
  Arms: Cervarix Group
Biological: Priorix — 1 dose administered intramuscularly in the deltoid muscle of the left arm at Day 0.
  Other Names: MMR
  Arms: Priorix + Infanrix Group
Biological: Infanrix — 1 dose administered intramuscularly in the deltoid muscle of the left arm at Month 6.
  Other Names: DTPa
  Arms: Priorix + Infanrix Group

SUMMARY:
The current study evaluates the immunogenicity and safety in 4-6 years old female subjects (experimental group) receiving Cervarix according to a 2-dose schedule (Month 0, 6), as compared to 4-6 years old female subjects (control group) receiving sequentially Priorix (Month 0) and Infanrix (Month 6) vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* A female between, and including, 4 and 6 years of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject prior to enrolment in the study.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects who received four doses of DTP vaccine (i.e., three doses in the first year of life and a fourth dose in the second year of life) according to the schedule applicable in the participating countries.
* Subjects who received a first dose of MMR vaccine according to the schedule applicable in the participating countries.

Exclusion Criteria:

* Child in care.
* Previous vaccination against HPV or planned administration of another HPV vaccine during the study other than that foreseen in the protocol.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of study vaccine(s). Administration of routine meningococcal, hepatitis B, hepatitis A, inactivated influenza and/or poliomyelitis vaccines up to 8 days before the first dose of study vaccine(s) is allowed. Enrolment will be deferred until the subject is outside of specified window.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine(s), or planned use during the study period.
* History of any reactions or hypersensitivity likely to be exacerbated by any component of the study vaccines, including latex and/or obvious allergic reactions to neomycin (a history of contact dermatitis to neomycin is not a contraindication), egg protein, etc. (e.g. hives, swelling of the mouth and throat, difficulty breathing, hypotension, or shock subsequent to egg ingestion).
* Cancer or autoimmune disease under treatment.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Previous administration of MPL or AS04 adjuvant.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine(s) or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* Documented human immunodeficiency virus (HIV)-positive subject.
* Major congenital defects or serious chronic illness.
* History of seizures or serious neurological disorder, which, according to the judgment of the investigator, precludes administration of any of the study vaccines.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests, which in the opinion of the investigator precludes administration of the study vaccine(s).
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 37.5°C on oral, axillary or tympanic setting, or ≥ 38.0°C on rectal setting.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator. Enrolment can be deferred until condition is resolved.
* Previous administration of the fifth dose of DTP vaccine and/or the second dose of MMR vaccine or planned administration of DTP vaccine and/or MMR vaccine outside the study (during the study period from Day 0 to Month 12).
* History of tetanus, diphtheria, pertussis, measles, mumps and/or rubella.
* Known exposure to diphtheria or household exposure to pertussis within 30 days prior to vaccination with DTPa.
* Known exposure to measles, mumps and/or rubella 30 days prior to vaccination with the MMR study vaccine.
* Confirmed or suspected tuberculosis.
* Severe allergic reactions (e.g. anaphylaxis or severe Arthus-type hypersensitivity reactions) following the administration of previous dose(s) of DTP or MMR vaccines.
* Hyperpyrexia (≥ 40.5°C) within 48 hours of administration of previous doses of DTP or MMR vaccines.
* Persistent, inconsolable crying lasting more than 3 hours, occurring within 48 hours of administration of previous doses of DTP vaccine.
* Collapse or shocking-like state (hypotonic-hyporesponsive episode) within 48 hours of administration of previous doses of DTP vaccine.
* Idiopathic thrombocytopenic purpura or bleeding disorders.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose(s). (For corticosteroids, this will mean prednisone ≥ 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.)

Ages: 4 Years to 6 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2012-10-15 (Actual); Primary Completion 2014-04-23 (Actual); Study Completion 2016-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Colombia (2):
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Yopal, Casanare
- GSK Investigational Site, México, Mexico
- GSK Investigational Site, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=16039

REFERENCES:
- [Background] Lin L, Parra MM, Sierra VY, Cespedes AS, Granados MA, Luque A, Damaso S, Castrejon Alba MM, Romano-Mazzotti L, Struyf F. Safety and Immunogenicity of the HPV-16/18 AS04-adjuvanted Vaccine in 4-6-year-old Girls: Results to Month 12 From a Randomized Trial. Pediatr Infect Dis J. 2018 Apr;37(4):e93-e102. doi: 10.1097/INF.0000000000001871. PMID 29424799
- [Background] Lin L, Macias Parra M, Sierra VY, Salas Cespedes A, Granados MA, Luque A, Karkada N, Castrejon Alba MM, Romano-Mazzotti L, Borys D, Struyf F. Long-term Immunogenicity and Safety of the AS04-adjuvanted Human Papillomavirus-16/18 Vaccine in Four- to Six-year-old Girls: Three-year Follow-up of a Randomized Phase III Trial. Pediatr Infect Dis J. 2019 Oct;38(10):1061-1067. doi: 10.1097/INF.0000000000002437. PMID 31469776
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted by multiple investigators at 7 centers in Colombia, Mexico and Panama.
Pre-assignment Details: All 148 subjects enrolled in the study, received the study vaccination and were included in the Total Vaccinated cohort (TVC).
Period: Overall Study
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Started | 74 | 74
Completed | 73 | 71
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Migrated/moved from study area | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Priorix + Infanrix Group | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.3 (0.5) | 4.4 (0.5) | 4.3 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 74 | 148
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage / African American | 4 | 2 | 6
  White - Caucasian / European Heritage | 2 | 4 | 6
  Mixed origin | 68 | 68 | 136

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 7-day follow-up period (i.e. from the day of vaccination up to 6 subsequent days) after each vaccine dose and across doses
Population: The analysis was based on the Total vaccinated cohort (TVC), which included all vaccinated subjects who received at least one dose of vaccine in this study, who had their symptom sheet filled in and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants
  Any Pain Dose 1 | 45 | 15
  Grade 3 Pain Dose 1 | 2 | 0
  Any Redness Dose 1 | 10 | 7
  Grade 3 Redness Dose 1 | 1 | 0
  Any Swelling Dose 1 | 6 | 6
  Grade 3 Swelling Dose 1 | 1 | 0
  Any Pain Dose 2: number analyzed (Participants) | 72 | 71
  Any Pain Dose 2 | 43 | 36
  Grade 3 Pain Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Pain Dose 2 | 2 | 1
  Any Redness Dose 2: number analyzed (Participants) | 72 | 71
  Any Redness Dose 2 | 12 | 12
  Grade 3 Redness Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Redness Dose 2 | 0 | 4
  Any Swelling Dose 2: number analyzed (Participants) | 72 | 71
  Any Swelling Dose 2 | 16 | 15
  Grade 3 Swelling Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Swelling Dose 2 | 3 | 7
  Any Pain Across doses | 54 | 40
  Grade 3 Pain Across doses | 4 | 1
  Any Redness Across doses | 18 | 18
  Grade 3 Redness Across doses | 1 | 4
  Any Swelling Across doses | 19 | 18
  Grade 3 Swelling Across doses | 4 | 7

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia (only in joints which were distal from the injection site), drowsiness, fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], gastrointestinal symptoms (nausea, vomiting, diarrhoea and/or abdominal pain), headache, irritability/fussiness, loss of appetite, myalgia, rash (not urticaria, not measels/rubella-like rash), urticaria. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Grade 3 irritability/fussiness = crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite = did not eat at all. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants
  Any Arthralgia Dose 1 | 5 | 8
  Grade 3 Arthralgia Dose 1 | 0 | 0
  Related Arthralgia Dose 1 | 4 | 8
  Any Drowsiness Dose 1 | 14 | 7
  Grade 3 Drowsiness Dose 1 | 3 | 0
  Related Drowsiness Dose 1 | 12 | 7
  Any Fatigue Dose 1 | 8 | 7
  Grade 3 Fatigue Dose 1 | 0 | 0
  Related Fatigue Dose 1 | 7 | 7
  Any Fever Dose 1 | 6 | 8
  Grade 3 Fever Dose 1 | 1 | 0
  Related Fever Dose 1 | 3 | 5
  Any Gastrointestinal Dose 1 | 7 | 12
  Grade 3 Gastrointestinal Dose 1 | 0 | 0
  Related Gastrointestinal Dose 1 | 5 | 10
  Any Headache Dose 1 | 11 | 19
  Grade 3 Headache Dose 1 | 0 | 1
  Related Headache Dose 1 | 9 | 17
  Any Irritability/fussiness Dose 1 | 13 | 7
  Grade 3 Irritability/fussiness Dose 1 | 1 | 0
  Related Irritability/fussiness Dose 1 | 12 | 7
  Any Loss of appetite Dose 1 | 15 | 7
  Grade 3 Loss of appetite Dose 1 | 0 | 0
  Related Loss of appetite Dose 1 | 13 | 7
  Any Myalgia Dose 1 | 13 | 9
  Grade 3 Myalgia Dose 1 | 0 | 0
  Related Myalgia Dose 1 | 13 | 9
  Any Rash Dose 1 | 3 | 1
  Grade 3 Rash Dose 1 | 0 | 0
  Related Rash Dose 1 | 2 | 1
  Any Urticaria Dose 1 | 5 | 3
  Grade 3 Urticaria Dose 1 | 0 | 0
  Related Urticaria Dose 1 | 4 | 3
  Any Arthralgia Dose 2: number analyzed (Participants) | 72 | 71
  Any Arthralgia Dose 2 | 10 | 8
  Grade 3 Arthralgia Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Arthralgia Dose 2 | 0 | 0
  Related Arthralgia Dose 2: number analyzed (Participants) | 72 | 71
  Related Arthralgia Dose 2 | 9 | 8
  Any Drowsiness Dose 2: number analyzed (Participants) | 72 | 71
  Any Drowsiness Dose 2 | 9 | 9
  Grade 3 Drowsiness Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Drowsiness Dose 2 | 0 | 0
  Related Drowsiness Dose 2: number analyzed (Participants) | 72 | 71
  Related Drowsiness Dose 2 | 9 | 9
  Any Fatigue Dose 2: number analyzed (Participants) | 72 | 71
  Any Fatigue Dose 2 | 9 | 7
  Grade 3 Fatigue Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Fatigue Dose 2 | 0 | 0
  Related Fatigue Dose 2: number analyzed (Participants) | 72 | 71
  Related Fatigue Dose 2 | 9 | 7
  Any Fever Dose 2: number analyzed (Participants) | 72 | 71
  Any Fever Dose 2 | 7 | 12
  Grade 3 Fever Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Fever Dose 2 | 0 | 0
  Related Fever Dose 2: number analyzed (Participants) | 72 | 71
  Related Fever Dose 2 | 7 | 9
  Any Gastrointestinal Dose 2: number analyzed (Participants) | 72 | 71
  Any Gastrointestinal Dose 2 | 4 | 9
  Grade 3 Gastrointestinal Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Gastrointestinal Dose 2 | 0 | 0
  Related Gastrointestinal Dose 2: number analyzed (Participants) | 72 | 71
  Related Gastrointestinal Dose 2 | 3 | 8
  Any Headache Dose 2: number analyzed (Participants) | 72 | 71
  Any Headache Dose 2 | 12 | 13
  Grade 3 Headache Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Headache Dose 2 | 0 | 0
  Related Headache Dose 2: number analyzed (Participants) | 72 | 71
  Related Headache Dose 2 | 12 | 12
  Any Irritability/fussiness Dose 2: number analyzed (Participants) | 72 | 71
  Any Irritability/fussiness Dose 2 | 18 | 17
  Grade 3 Irritability/fussiness Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Irritability/fussiness Dose 2 | 0 | 0
  Related Irritability/fussiness Dose 2: number analyzed (Participants) | 72 | 71
  Related Irritability/fussiness Dose 2 | 18 | 17
  Any Loss of appetite Dose 2: number analyzed (Participants) | 72 | 71
  Any Loss of appetite Dose 2 | 9 | 8
  Grade 3 Loss of appetite Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Loss of appetite Dose 2 | 1 | 1
  Related Loss of appetite Dose 2: number analyzed (Participants) | 72 | 71
  Related Loss of appetite Dose 2 | 9 | 8
  Any Myalgia Dose 2: number analyzed (Participants) | 72 | 71
  Any Myalgia Dose 2 | 13 | 11
  Grade 3 Myalgia Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Myalgia Dose 2 | 0 | 0
  Related Myalgia Dose 2: number analyzed (Participants) | 72 | 71
  Related Myalgia Dose 2 | 12 | 11
  Any Rash Dose 2: number analyzed (Participants) | 72 | 71
  Any Rash Dose 2 | 3 | 4
  Grade 3 Rash Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Rash Dose 2 | 0 | 0
  Related Rash Dose 2: number analyzed (Participants) | 72 | 71
  Related Rash Dose 2 | 3 | 3
  Any Urticaria Dose 2: number analyzed (Participants) | 72 | 71
  Any Urticaria Dose 2 | 5 | 4
  Grade 3 Urticaria Dose 2: number analyzed (Participants) | 72 | 71
  Grade 3 Urticaria Dose 2 | 0 | 0
  Related Urticaria Dose 2: number analyzed (Participants) | 72 | 71
  Related Urticaria Dose 2 | 4 | 3
  Any Arthralgia Across doses | 13 | 11
  Grade 3 Arthralgia Across doses | 0 | 0
  Related Arthralgia Across doses | 12 | 11
  Any Drowsiness Across doses | 16 | 15
  Grade 3 Drowsiness Across doses | 3 | 0
  Related Drowsiness Across doses | 15 | 15
  Any Fatigue Across doses | 15 | 10
  Grade 3 Fatigue Across doses | 0 | 0
  Related Fatigue Across doses | 14 | 10
  Any Fever Across doses | 12 | 17
  Grade 3 Fever Across doses | 1 | 0
  Related Fever Across doses | 9 | 13
  Any Gastrointestinal Across doses | 11 | 16
  Grade 3 Gastrointestinal Across doses | 0 | 0
  Related Gastrointestinal Across doses | 8 | 15
  Any Headache Across doses | 18 | 25
  Grade 3 Headache Across doses | 0 | 1
  Related Headache Across doses | 16 | 23
  Any Irritability/fussiness Across doses | 22 | 19
  Grade 3 Irritability/fussiness Across doses | 1 | 0
  Related Irritability/fussiness Across doses | 22 | 19
  Any Loss of appetite Across doses | 21 | 13
  Grade 3 Loss of appetite Across doses | 1 | 1
  Related Loss of appetite Across doses | 19 | 13
  Any Myalgia Across doses | 21 | 14
  Grade 3 Myalgia Across doses | 0 | 0
  Related Myalgia Across doses | 21 | 14
  Any Rash Across doses | 6 | 5
  Grade 3 Rash Across doses | 0 | 0
  Related Rash Across doses | 5 | 4
  Any Urticaria Across doses | 10 | 7
  Grade 3 Urticaria Across doses | 0 | 0
  Related Urticaria Across doses | 8 | 6

3. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs) Reported During the 43-day Period Following the Vaccination at Day 0
Description: An unsolicited AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also included failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related AE = AE assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 43-day period (i.e. from the day of vaccination up to 42 subsequent days) following the vaccination at Day 0
Population: The analysis was based on the Total vaccinated cohort (TVC), which included all vaccinated subjects who received at least one dose of vaccine in this study and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants
  Any AE(s) | 40 | 40
  Grade 3 AE(s) | 3 | 2
  Related AE(s) | 1 | 5

4. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited AEs Reported During the 30-day Period Following the Vaccination at Month 6
Description: as for outcome 3
Time Frame: During the 30-day period (i.e. from the day of vaccination up to 29 subsequent days) following the vaccination at Month 6
Population: The analysis was based on the Total vaccinated cohort (TVC), which included all vaccinated subjects who received at least one dose of vaccine in this study and for whom data were available. Out of the 74 subjects present in the initial Priorix + Infanrix Group, 3 did not receive the second vaccination and were hence excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 71
Participants
  Any AE(s) | 18 | 13
  Grade 3 AE(s) | 0 | 0
  Related AE(s) | 0 | 1

5. Primary Outcome: Number of Subjects With Clinically Relevant Abnormalities in Biochemical and Haematological Parameters at Day 42 by Baseline Ranges
Description: The parameters assessed were both biochemical (alanine aminotransferase = ALAT, creatinine = CREA, blood urea nitrogen = BUN) and haematological (basophils = BAS, eosinophils = EOS, red blood cells = RBC, hematocrit = HCT, hemoglobin = HGB, leukocytes [white blood cells] = WBC, lymphocytes = LYM, monocytes = MONO, neutrophils = NEU and platelets = PLA).
  Abnormal laboratory values at Day 42 were Below, Within and Above normal ranges, as compared to the baseline status of the same parameter, at Day 0 (Unknown, Below, Within and Above normal ranges) [e.g. ALAT Below (baseline) - Within (Day 42) = ALAT with below normal value at baseline and within normal values at Day 42].
Time Frame: At Day 42 (i.e. 42 days after the vaccination at Day 0)
Population: The analysis was based on the Total vaccinated cohort (TVC), which included all vaccinated subjects who received at least one dose of vaccine in this study and for whom data were available at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 73
Participants
  ALAT, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 2 | 2
  ALAT, Unknown (baseline) - Below (Day 42) | 0 | 0
  ALAT, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 2 | 2
  ALAT, Unknown (baseline) - Within (Day 42) | 2 | 1
  ALAT, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 2 | 2
  ALAT, Unknown (baseline) - Above (Day 42) | 0 | 1
  ALAT, Below (baseline) - Below (Day 42): number analyzed (Participants) | 2 | 1
  ALAT, Below (baseline) - Below (Day 42) | 1 | 0
  ALAT, Below (baseline) - Within (Day 42): number analyzed (Participants) | 2 | 1
  ALAT, Below (baseline) - Within (Day 42) | 1 | 1
  ALAT, Below (baseline) - Above (Day 42): number analyzed (Participants) | 2 | 1
  ALAT, Below (baseline) - Above (Day 42) | 0 | 0
  ALAT, Within (baseline) - Below (Day 42): number analyzed (Participants) | 66 | 62
  ALAT, Within (baseline) - Below (Day 42) | 0 | 0
  ALAT, Within (baseline) - Within (Day 42): number analyzed (Participants) | 66 | 62
  ALAT, Within (baseline) - Within (Day 42) | 64 | 60
  ALAT, Within (baseline) - Above (Day 42): number analyzed (Participants) | 66 | 62
  ALAT, Within (baseline) - Above (Day 42) | 2 | 2
  ALAT, Above (baseline) - Below (Day 42): number analyzed (Participants) | 4 | 7
  ALAT, Above (baseline) - Below (Day 42) | 0 | 0
  ALAT, Above (baseline) - Within (Day 42): number analyzed (Participants) | 4 | 7
  ALAT, Above (baseline) - Within (Day 42) | 1 | 4
  ALAT, Above (baseline) - Above (Day 42): number analyzed (Participants) | 4 | 7
  ALAT, Above (baseline) - Above (Day 42) | 3 | 3
  BAS, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 1 | 0
  BAS, Unknown (baseline) - Below (Day 42) | 0 |
  BAS, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 1 | 0
  BAS, Unknown (baseline) - Within (Day 42) | 1 |
  BAS, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 1 | 0
  BAS, Unknown (baseline) - Above (Day 42) | 0 |
  BAS, Below (baseline) - Below (Day 42): number analyzed (Participants) | 0 | 0
  BAS, Below (baseline) - Within (Day 42): number analyzed (Participants) | 0 | 0
  BAS, Below (baseline) - Above (Day 42): number analyzed (Participants) | 0 | 0
  BAS, Within (baseline) - Below (Day 42): number analyzed (Participants) | 71 | 69
  BAS, Within (baseline) - Below (Day 42) | 0 | 0
  BAS, Within (baseline) - Within (Day 42): number analyzed (Participants) | 71 | 69
  BAS, Within (baseline) - Within (Day 42) | 71 | 69
  BAS, Within (baseline) - Above (Day 42): number analyzed (Participants) | 71 | 69
  BAS, Within (baseline) - Above (Day 42) | 0 | 0
  BAS, Above (baseline) - Below (Day 42): number analyzed (Participants) | 0 | 4
  BAS, Above (baseline) - Below (Day 42) |  | 0
  BAS, Above (baseline) - Within (Day 42): number analyzed (Participants) | 0 | 4
  BAS, Above (baseline) - Within (Day 42) |  | 4
  BAS, Above (baseline) - Above (Day 42): number analyzed (Participants) | 0 | 4
  BAS, Above (baseline) - Above (Day 42) |  | 0
  CREA, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 2 | 1
  CREA, Unknown (baseline) - Below (Day 42) | 0 | 1
  CREA, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 2 | 1
  CREA, Unknown (baseline) - Within (Day 42) | 2 | 0
  CREA, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 2 | 1
  CREA, Unknown (baseline) - Above (Day 42) | 0 | 0
  CREA, Below (baseline) - Below (Day 42): number analyzed (Participants) | 30 | 27
  CREA, Below (baseline) - Below (Day 42) | 22 | 17
  CREA, Below (baseline) - Within (Day 42): number analyzed (Participants) | 30 | 27
  CREA, Below (baseline) - Within (Day 42) | 8 | 10
  CREA, Below (baseline) - Above (Day 42): number analyzed (Participants) | 30 | 27
  CREA, Below (baseline) - Above (Day 42) | 0 | 0
  CREA, Within (baseline) - Below (Day 42): number analyzed (Participants) | 42 | 45
  CREA, Within (baseline) - Below (Day 42) | 7 | 12
  CREA, Within (baseline) - Within (Day 42): number analyzed (Participants) | 42 | 45
  CREA, Within (baseline) - Within (Day 42) | 35 | 33
  CREA, Within (baseline) - Above (Day 42): number analyzed (Participants) | 42 | 45
  CREA, Within (baseline) - Above (Day 42) | 0 | 0
  CREA, Above (baseline) - Below (Day 42): number analyzed (Participants) | 0 | 0
  CREA, Above (baseline) - Within (Day 42): number analyzed (Participants) | 0 | 0
  CREA, Above (baseline) - Above (Day 42): number analyzed (Participants) | 0 | 0
  EOS, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 1 | 0
  EOS, Unknown (baseline) - Below (Day 42) | 0 |
  EOS, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 1 | 0
  EOS, Unknown (baseline) - Within (Day 42) | 1 |
  EOS, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 1 | 0
  EOS, Unknown (baseline) - Above (Day 42) | 0 |
  EOS, Below (baseline) - Below (Day 42): number analyzed (Participants) | 1 | 0
  EOS, Below (baseline) - Below (Day 42) | 0 |
  EOS, Below (baseline) - Within (Day 42): number analyzed (Participants) | 1 | 0
  EOS, Below (baseline) - Within (Day 42) | 1 |
  EOS, Below (baseline) - Above (Day 42): number analyzed (Participants) | 1 | 0
  EOS, Below (baseline) - Above (Day 42) | 0 |
  EOS, Within (baseline) - Below (Day 42): number analyzed (Participants) | 49 | 50
  EOS, Within (baseline) - Below (Day 42) | 1 | 1
  EOS, Within (baseline) - Within (Day 42): number analyzed (Participants) | 49 | 50
  EOS, Within (baseline) - Within (Day 42) | 42 | 38
  EOS, Within (baseline) - Above (Day 42): number analyzed (Participants) | 49 | 50
  EOS, Within (baseline) - Above (Day 42) | 6 | 11
  EOS, Above (baseline) - Below (Day 42): number analyzed (Participants) | 21 | 23
  EOS, Above (baseline) - Below (Day 42) | 0 | 1
  EOS, Above (baseline) - Within (Day 42): number analyzed (Participants) | 21 | 23
  EOS, Above (baseline) - Within (Day 42) | 4 | 10
  EOS, Above (baseline) - Above (Day 42): number analyzed (Participants) | 21 | 23
  EOS, Above (baseline) - Above (Day 42) | 17 | 12
  RBC, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 1 | 0
  RBC, Unknown (baseline) - Below (Day 42) | 0 |
  RBC, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 1 | 0
  RBC, Unknown (baseline) - Within (Day 42) | 1 |
  RBC, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 1 | 0
  RBC, Unknown (baseline) - Above (Day 42) | 0 |
  RBC, Below (baseline) - Below (Day 42): number analyzed (Participants) | 5 | 5
  RBC, Below (baseline) - Below (Day 42) | 0 | 1
  RBC, Below (baseline) - Within (Day 42): number analyzed (Participants) | 5 | 5
  RBC, Below (baseline) - Within (Day 42) | 5 | 4
  RBC, Below (baseline) - Above (Day 42): number analyzed (Participants) | 5 | 5
  RBC, Below (baseline) - Above (Day 42) | 0 | 0
  RBC, Within (baseline) - Below (Day 42): number analyzed (Participants) | 66 | 66
  RBC, Within (baseline) - Below (Day 42) | 5 | 2
  RBC, Within (baseline) - Within (Day 42): number analyzed (Participants) | 66 | 66
  RBC, Within (baseline) - Within (Day 42) | 60 | 63
  RBC, Within (baseline) - Above (Day 42): number analyzed (Participants) | 66 | 66
  RBC, Within (baseline) - Above (Day 42) | 1 | 1
  RBC, Above (baseline) - Below (Day 42): number analyzed (Participants) | 0 | 2
  RBC, Above (baseline) - Below (Day 42) |  | 0
  RBC, Above (baseline) - Within (Day 42): number analyzed (Participants) | 0 | 2
  RBC, Above (baseline) - Within (Day 42) |  | 1
  RBC, Above (baseline) - Above (Day 42): number analyzed (Participants) | 0 | 2
  RBC, Above (baseline) - Above (Day 42) |  | 1
  HCT, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 1 | 0
  HCT, Unknown (baseline) - Below (Day 42) | 0 |
  HCT, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 1 | 0
  HCT, Unknown (baseline) - Within (Day 42) | 1 |
  HCT, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 1 | 0
  HCT, Unknown (baseline) - Above (Day 42) | 0 |
  HCT, Below (baseline) - Below (Day 42): number analyzed (Participants) | 25 | 24
  HCT, Below (baseline) - Below (Day 42) | 12 | 15
  HCT, Below (baseline) - Within (Day 42): number analyzed (Participants) | 25 | 24
  HCT, Below (baseline) - Within (Day 42) | 13 | 8
  HCT, Below (baseline) - Above (Day 42): number analyzed (Participants) | 25 | 24
  HCT, Below (baseline) - Above (Day 42) | 0 | 1
  HCT, Within (baseline) - Below (Day 42): number analyzed (Participants) | 43 | 45
  HCT, Within (baseline) - Below (Day 42) | 5 | 2
  HCT, Within (baseline) - Within (Day 42): number analyzed (Participants) | 43 | 45
  HCT, Within (baseline) - Within (Day 42) | 37 | 38
  HCT, Within (baseline) - Above (Day 42): number analyzed (Participants) | 43 | 45
  HCT, Within (baseline) - Above (Day 42) | 1 | 5
  HCT, Above (baseline) - Below (Day 42): number analyzed (Participants) | 3 | 4
  HCT, Above (baseline) - Below (Day 42) | 0 | 0
  HCT, Above (baseline) - Within (Day 42): number analyzed (Participants) | 3 | 4
  HCT, Above (baseline) - Within (Day 42) | 2 | 4
  HCT, Above (baseline) - Above (Day 42): number analyzed (Participants) | 3 | 4
  HCT, Above (baseline) - Above (Day 42) | 1 | 0
  HGB, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 1 | 0
  HGB, Unknown (baseline) - Below (Day 42) | 0 |
  HGB, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 1 | 0
  HGB, Unknown (baseline) - Within (Day 42) | 0 |
  HGB, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 1 | 0
  HGB, Unknown (baseline) - Above (Day 42) | 1 |
  HGB, Below (baseline) - Below (Day 42): number analyzed (Participants) | 20 | 14
  HGB, Below (baseline) - Below (Day 42) | 10 | 5
  HGB, Below (baseline) - Within (Day 42): number analyzed (Participants) | 20 | 14
  HGB, Below (baseline) - Within (Day 42) | 10 | 9
  HGB, Below (baseline) - Above (Day 42): number analyzed (Participants) | 20 | 14
  HGB, Below (baseline) - Above (Day 42) | 0 | 0
  HGB, Within (baseline) - Below (Day 42): number analyzed (Participants) | 46 | 53
  HGB, Within (baseline) - Below (Day 42) | 4 | 7
  HGB, Within (baseline) - Within (Day 42): number analyzed (Participants) | 46 | 53
  HGB, Within (baseline) - Within (Day 42) | 38 | 42
  HGB, Within (baseline) - Above (Day 42): number analyzed (Participants) | 46 | 53
  HGB, Within (baseline) - Above (Day 42) | 4 | 4
  HGB, Above (baseline) - Below (Day 42): number analyzed (Participants) | 5 | 6
  HGB, Above (baseline) - Below (Day 42) | 0 | 0
  HGB, Above (baseline) - Within (Day 42): number analyzed (Participants) | 5 | 6
  HGB, Above (baseline) - Within (Day 42) | 3 | 5
  HGB, Above (baseline) - Above (Day 42): number analyzed (Participants) | 5 | 6
  HGB, Above (baseline) - Above (Day 42) | 2 | 1
  WBC, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 1 | 0
  WBC, Unknown (baseline) - Below (Day 42) | 0 |
  WBC, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 1 | 0
  WBC, Unknown (baseline) - Within (Day 42) | 1 |
  WBC, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 1 | 0
  WBC, Unknown (baseline) - Above (Day 42) | 0 |
  WBC, Below (baseline) - Below (Day 42): number analyzed (Participants) | 5 | 7
  WBC, Below (baseline) - Below (Day 42) | 1 | 5
  WBC, Below (baseline) - Within (Day 42): number analyzed (Participants) | 5 | 7
  WBC, Below (baseline) - Within (Day 42) | 3 | 1
  WBC, Below (baseline) - Above (Day 42): number analyzed (Participants) | 5 | 7
  WBC, Below (baseline) - Above (Day 42) | 1 | 1
  WBC, Within (baseline) - Below (Day 42): number analyzed (Participants) | 62 | 59
  WBC, Within (baseline) - Below (Day 42) | 2 | 1
  WBC, Within (baseline) - Within (Day 42): number analyzed (Participants) | 62 | 59
  WBC, Within (baseline) - Within (Day 42) | 57 | 54
  WBC, Within (baseline) - Above (Day 42): number analyzed (Participants) | 62 | 59
  WBC, Within (baseline) - Above (Day 42) | 3 | 4
  WBC, Above (baseline) - Below (Day 42): number analyzed (Participants) | 4 | 7
  WBC, Above (baseline) - Below (Day 42) | 0 | 0
  WBC, Above (baseline) - Within (Day 42): number analyzed (Participants) | 4 | 7
  WBC, Above (baseline) - Within (Day 42) | 1 | 4
  WBC, Above (baseline) - Above (Day 42): number analyzed (Participants) | 4 | 7
  WBC, Above (baseline) - Above (Day 42) | 3 | 3
  LYM, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 1 | 0
  LYM, Unknown (baseline) - Below (Day 42) | 0 |
  LYM, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 1 | 0
  LYM, Unknown (baseline) - Within (Day 42) | 1 |
  LYM, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 1 | 0
  LYM, Unknown (baseline) - Above (Day 42) | 0 |
  LYM, Below (baseline) - Below (Day 42): number analyzed (Participants) | 7 | 10
  LYM, Below (baseline) - Below (Day 42) | 4 | 6
  LYM, Below (baseline) - Within (Day 42): number analyzed (Participants) | 7 | 10
  LYM, Below (baseline) - Within (Day 42) | 2 | 2
  LYM, Below (baseline) - Above (Day 42): number analyzed (Participants) | 7 | 10
  LYM, Below (baseline) - Above (Day 42) | 1 | 2
  LYM, Within (baseline) - Below (Day 42): number analyzed (Participants) | 48 | 42
  LYM, Within (baseline) - Below (Day 42) | 7 | 2
  LYM, Within (baseline) - Within (Day 42): number analyzed (Participants) | 48 | 42
  LYM, Within (baseline) - Within (Day 42) | 38 | 34
  LYM, Within (baseline) - Above (Day 42): number analyzed (Participants) | 48 | 42
  LYM, Within (baseline) - Above (Day 42) | 3 | 6
  LYM, Above (baseline) - Below (Day 42): number analyzed (Participants) | 16 | 21
  LYM, Above (baseline) - Below (Day 42) | 0 | 2
  LYM, Above (baseline) - Within (Day 42): number analyzed (Participants) | 16 | 21
  LYM, Above (baseline) - Within (Day 42) | 5 | 5
  LYM, Above (baseline) - Above (Day 42): number analyzed (Participants) | 16 | 21
  LYM, Above (baseline) - Above (Day 42) | 11 | 14
  MONO, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 1 | 0
  MONO, Unknown (baseline) - Below (Day 42) | 1 |
  MONO, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 1 | 0
  MONO, Unknown (baseline) - Within (Day 42) | 0 |
  MONO, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 1 | 0
  MONO, Unknown (baseline) - Above (Day 42) | 0 |
  MONO, Below (baseline) - Below (Day 42): number analyzed (Participants) | 8 | 9
  MONO, Below (baseline) - Below (Day 42) | 4 | 5
  MONO, Below (baseline) - Within (Day 42): number analyzed (Participants) | 8 | 9
  MONO, Below (baseline) - Within (Day 42) | 4 | 4
  MONO, Below (baseline) - Above (Day 42): number analyzed (Participants) | 8 | 9
  MONO, Below (baseline) - Above (Day 42) | 0 | 0
  MONO, Within (baseline) - Below (Day 42): number analyzed (Participants) | 51 | 55
  MONO, Within (baseline) - Below (Day 42) | 3 | 2
  MONO, Within (baseline) - Within (Day 42): number analyzed (Participants) | 51 | 55
  MONO, Within (baseline) - Within (Day 42) | 42 | 48
  MONO, Within (baseline) - Above (Day 42): number analyzed (Participants) | 51 | 55
  MONO, Within (baseline) - Above (Day 42) | 6 | 5
  MONO, Above (baseline) - Below (Day 42): number analyzed (Participants) | 12 | 9
  MONO, Above (baseline) - Below (Day 42) | 0 | 0
  MONO, Above (baseline) - Within (Day 42): number analyzed (Participants) | 12 | 9
  MONO, Above (baseline) - Within (Day 42) | 6 | 3
  MONO, Above (baseline) - Above (Day 42): number analyzed (Participants) | 12 | 9
  MONO, Above (baseline) - Above (Day 42) | 6 | 6
  NEU, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 1 | 0
  NEU, Unknown (baseline) - Below (Day 42) | 0 |
  NEU, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 1 | 0
  NEU, Unknown (baseline) - Within (Day 42) | 1 |
  NEU, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 1 | 0
  NEU, Unknown (baseline) - Above (Day 42) | 0 |
  NEU, Below (baseline) - Below (Day 42): number analyzed (Participants) | 15 | 21
  NEU, Below (baseline) - Below (Day 42) | 9 | 14
  NEU, Below (baseline) - Within (Day 42): number analyzed (Participants) | 15 | 21
  NEU, Below (baseline) - Within (Day 42) | 6 | 6
  NEU, Below (baseline) - Above (Day 42): number analyzed (Participants) | 15 | 21
  NEU, Below (baseline) - Above (Day 42) | 0 | 1
  NEU, Within (baseline) - Below (Day 42): number analyzed (Participants) | 52 | 46
  NEU, Within (baseline) - Below (Day 42) | 4 | 6
  NEU, Within (baseline) - Within (Day 42): number analyzed (Participants) | 52 | 46
  NEU, Within (baseline) - Within (Day 42) | 41 | 39
  NEU, Within (baseline) - Above (Day 42): number analyzed (Participants) | 52 | 46
  NEU, Within (baseline) - Above (Day 42) | 7 | 1
  NEU, Above (baseline) - Below (Day 42): number analyzed (Participants) | 4 | 6
  NEU, Above (baseline) - Below (Day 42) | 0 | 0
  NEU, Above (baseline) - Within (Day 42): number analyzed (Participants) | 4 | 6
  NEU, Above (baseline) - Within (Day 42) | 3 | 3
  NEU, Above (baseline) - Above (Day 42): number analyzed (Participants) | 4 | 6
  NEU, Above (baseline) - Above (Day 42) | 1 | 3
  PLA, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 2 | 0
  PLA, Unknown (baseline) - Below (Day 42) | 0 |
  PLA, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 2 | 0
  PLA, Unknown (baseline) - Within (Day 42) | 2 |
  PLA, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 2 | 0
  PLA, Unknown (baseline) - Above (Day 42) | 0 |
  PLA, Below (baseline) - Below (Day 42): number analyzed (Participants) | 0 | 2
  PLA, Below (baseline) - Below (Day 42) |  | 0
  PLA, Below (baseline) - Within (Day 42): number analyzed (Participants) | 0 | 2
  PLA, Below (baseline) - Within (Day 42) |  | 2
  PLA, Below (baseline) - Above (Day 42): number analyzed (Participants) | 0 | 2
  PLA, Below (baseline) - Above (Day 42) |  | 0
  PLA, Within (baseline) - Below (Day 42): number analyzed (Participants) | 59 | 56
  PLA, Within (baseline) - Below (Day 42) | 0 | 0
  PLA, Within (baseline) - Within (Day 42): number analyzed (Participants) | 59 | 56
  PLA, Within (baseline) - Within (Day 42) | 51 | 52
  PLA, Within (baseline) - Above (Day 42): number analyzed (Participants) | 59 | 56
  PLA, Within (baseline) - Above (Day 42) | 8 | 4
  PLA, Above (baseline) - Below (Day 42): number analyzed (Participants) | 11 | 15
  PLA, Above (baseline) - Below (Day 42) | 0 | 0
  PLA, Above (baseline) - Within (Day 42): number analyzed (Participants) | 11 | 15
  PLA, Above (baseline) - Within (Day 42) | 4 | 9
  PLA, Above (baseline) - Above (Day 42): number analyzed (Participants) | 11 | 15
  PLA, Above (baseline) - Above (Day 42) | 7 | 6
  BUN, Unknown (baseline) - Below (Day 42): number analyzed (Participants) | 2 | 1
  BUN, Unknown (baseline) - Below (Day 42) | 0 | 0
  BUN, Unknown (baseline) - Within (Day 42): number analyzed (Participants) | 2 | 1
  BUN, Unknown (baseline) - Within (Day 42) | 2 | 1
  BUN, Unknown (baseline) - Above (Day 42): number analyzed (Participants) | 2 | 1
  BUN, Unknown (baseline) - Above (Day 42) | 0 | 0
  BUN, Below (baseline) - Below (Day 42): number analyzed (Participants) | 12 | 4
  BUN, Below (baseline) - Below (Day 42) | 4 | 1
  BUN, Below (baseline) - Within (Day 42): number analyzed (Participants) | 12 | 4
  BUN, Below (baseline) - Within (Day 42) | 8 | 3
  BUN, Below (baseline) - Above (Day 42): number analyzed (Participants) | 12 | 4
  BUN, Below (baseline) - Above (Day 42) | 0 | 0
  BUN, Within (baseline) - Below (Day 42): number analyzed (Participants) | 54 | 62
  BUN, Within (baseline) - Below (Day 42) | 2 | 5
  BUN, Within (baseline) - Within (Day 42): number analyzed (Participants) | 54 | 62
  BUN, Within (baseline) - Within (Day 42) | 50 | 57
  BUN, Within (baseline) - Above (Day 42): number analyzed (Participants) | 54 | 62
  BUN, Within (baseline) - Above (Day 42) | 2 | 0
  BUN, Above (baseline) - Below (Day 42): number analyzed (Participants) | 6 | 6
  BUN, Above (baseline) - Below (Day 42) | 0 | 0
  BUN, Above (baseline) - Within (Day 42): number analyzed (Participants) | 6 | 6
  BUN, Above (baseline) - Within (Day 42) | 6 | 6
  BUN, Above (baseline) - Above (Day 42): number analyzed (Participants) | 6 | 6
  BUN, Above (baseline) - Above (Day 42) | 0 | 0

6. Primary Outcome: Number of Subjects With Clinically Relevant Abnormalities in Biochemical and Haematological Parameters at Month 7 by Baseline Ranges
Description: The parameters assessed were both biochemical (alanine aminotransferase = ALAT, creatinine = CREA, blood urea nitrogen = BUN) and haematological (basophils = BAS, eosinophils = EOS, red blood cells = RBC, hematocrit = HCT, hemoglobin = HGB, leukocytes [white blood cells] = WBC, lymphocytes = LYM, monocytes = MONO, neutrophils = NEU and platelets = PLA). Abnormal laboratory values at Month 7 were Below, Within and Above normal ranges, as compared to the baseline status of the same parameter, at Day 0 (Unknown, Below, Within and Above normal ranges) [e.g. ALAT Below (baseline) - Within (Month 7) = ALAT with below normal value at baseline and within normal values at Month 7].
Time Frame: At Month 7 (i.e. 30 days after the vaccination at Month 6)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 72
Participants
  ALAT, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 2 | 2
  ALAT, Unknown (baseline) - Below (Month 7) | 0 | 0
  ALAT, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 2 | 2
  ALAT, Unknown (baseline) - Within (Month 7) | 2 | 2
  ALAT, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 2 | 2
  ALAT, Unknown (baseline) - Above (Month 7) | 0 | 0
  ALAT, Below (baseline) - Below (Month 7): number analyzed (Participants) | 2 | 1
  ALAT, Below (baseline) - Below (Month 7) | 1 | 0
  ALAT, Below (baseline) - Within (Month 7): number analyzed (Participants) | 2 | 1
  ALAT, Below (baseline) - Within (Month 7) | 1 | 1
  ALAT, Below (baseline) - Above (Month 7): number analyzed (Participants) | 2 | 1
  ALAT, Below (baseline) - Above (Month 7) | 0 | 0
  ALAT, Within (baseline) - Below (Month 7): number analyzed (Participants) | 65 | 62
  ALAT, Within (baseline) - Below (Month 7) | 1 | 1
  ALAT, Within (baseline) - Within (Month 7): number analyzed (Participants) | 65 | 62
  ALAT, Within (baseline) - Within (Month 7) | 64 | 60
  ALAT, Within (baseline) - Above (Month 7): number analyzed (Participants) | 65 | 62
  ALAT, Within (baseline) - Above (Month 7) | 0 | 1
  ALAT, Above (baseline) - Below (Month 7): number analyzed (Participants) | 4 | 7
  ALAT, Above (baseline) - Below (Month 7) | 0 | 0
  ALAT, Above (baseline) - Within (Month 7): number analyzed (Participants) | 4 | 7
  ALAT, Above (baseline) - Within (Month 7) | 3 | 7
  ALAT, Above (baseline) - Above (Month 7): number analyzed (Participants) | 4 | 7
  ALAT, Above (baseline) - Above (Month 7) | 1 | 0
  BAS, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 1 | 0
  BAS, Unknown (baseline) - Below (Month 7) | 0 |
  BAS, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 1 | 0
  BAS, Unknown (baseline) - Within (Month 7) | 1 |
  BAS, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 1 | 0
  BAS, Unknown (baseline) - Above (Month 7) | 0 |
  BAS, Below (baseline) - Below (Month 7): number analyzed (Participants) | 0 | 0
  BAS, Below (baseline) - Within (Month 7): number analyzed (Participants) | 0 | 0
  BAS, Below (baseline) - Above (Month 7): number analyzed (Participants) | 0 | 0
  BAS, Within (baseline) - Below (Month 7): number analyzed (Participants) | 73 | 68
  BAS, Within (baseline) - Below (Month 7) | 0 | 0
  BAS, Within (baseline) - Within (Month 7): number analyzed (Participants) | 73 | 68
  BAS, Within (baseline) - Within (Month 7) | 72 | 67
  BAS, Within (baseline) - Above (Month 7): number analyzed (Participants) | 73 | 68
  BAS, Within (baseline) - Above (Month 7) | 1 | 1
  BAS, Above (baseline) - Below (Month 7): number analyzed (Participants) | 0 | 4
  BAS, Above (baseline) - Below (Month 7) |  | 0
  BAS, Above (baseline) - Within (Month 7): number analyzed (Participants) | 0 | 4
  BAS, Above (baseline) - Within (Month 7) |  | 2
  BAS, Above (baseline) - Above (Month 7): number analyzed (Participants) | 0 | 4
  BAS, Above (baseline) - Above (Month 7) |  | 2
  CREA, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 2 | 1
  CREA, Unknown (baseline) - Below (Month 7) | 1 | 1
  CREA, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 2 | 1
  CREA, Unknown (baseline) - Within (Month 7) | 1 | 0
  CREA, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 2 | 1
  CREA, Unknown (baseline) - Above (Month 7) | 0 | 0
  CREA, Below (baseline) - Below (Month 7): number analyzed (Participants) | 29 | 26
  CREA, Below (baseline) - Below (Month 7) | 23 | 21
  CREA, Below (baseline) - Within (Month 7): number analyzed (Participants) | 29 | 26
  CREA, Below (baseline) - Within (Month 7) | 6 | 5
  CREA, Below (baseline) - Above (Month 7): number analyzed (Participants) | 29 | 26
  CREA, Below (baseline) - Above (Month 7) | 0 | 0
  CREA, Within (baseline) - Below (Month 7): number analyzed (Participants) | 42 | 45
  CREA, Within (baseline) - Below (Month 7) | 8 | 9
  CREA, Within (baseline) - Within (Month 7): number analyzed (Participants) | 42 | 45
  CREA, Within (baseline) - Within (Month 7) | 34 | 36
  CREA, Within (baseline) - Above (Month 7): number analyzed (Participants) | 42 | 45
  CREA, Within (baseline) - Above (Month 7) | 0 | 0
  CREA, Above (baseline) - Below (Month 7): number analyzed (Participants) | 0 | 0
  CREA, Above (baseline) - Within (Month 7): number analyzed (Participants) | 0 | 0
  CREA, Above (baseline) - Above (Month 7): number analyzed (Participants) | 0 | 0
  EOS, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 1 | 0
  EOS, Unknown (baseline) - Below (Month 7) | 0 |
  EOS, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 1 | 0
  EOS, Unknown (baseline) - Within (Month 7) | 1 |
  EOS, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 1 | 0
  EOS, Unknown (baseline) - Above (Month 7) | 0 |
  EOS, Below (baseline) - Below (Month 7): number analyzed (Participants) | 1 | 0
  EOS, Below (baseline) - Below (Month 7) | 0 |
  EOS, Below (baseline) - Within (Month 7): number analyzed (Participants) | 1 | 0
  EOS, Below (baseline) - Within (Month 7) | 1 |
  EOS, Below (baseline) - Above (Month 7): number analyzed (Participants) | 1 | 0
  EOS, Below (baseline) - Above (Month 7) | 0 |
  EOS, Within (baseline) - Below (Month 7): number analyzed (Participants) | 51 | 49
  EOS, Within (baseline) - Below (Month 7) | 0 | 1
  EOS, Within (baseline) - Within (Month 7): number analyzed (Participants) | 51 | 49
  EOS, Within (baseline) - Within (Month 7) | 42 | 38
  EOS, Within (baseline) - Above (Month 7): number analyzed (Participants) | 51 | 49
  EOS, Within (baseline) - Above (Month 7) | 9 | 10
  EOS, Above (baseline) - Below (Month 7): number analyzed (Participants) | 21 | 23
  EOS, Above (baseline) - Below (Month 7) | 0 | 0
  EOS, Above (baseline) - Within (Month 7): number analyzed (Participants) | 21 | 23
  EOS, Above (baseline) - Within (Month 7) | 3 | 10
  EOS, Above (baseline) - Above (Month 7): number analyzed (Participants) | 21 | 23
  EOS, Above (baseline) - Above (Month 7) | 18 | 13
  RBC, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 1 | 0
  RBC, Unknown (baseline) - Below (Month 7) | 0 |
  RBC, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 1 | 0
  RBC, Unknown (baseline) - Within (Month 7) | 1 |
  RBC, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 1 | 0
  RBC, Unknown (baseline) - Above (Month 7) | 0 |
  RBC, Below (baseline) - Below (Month 7): number analyzed (Participants) | 5 | 5
  RBC, Below (baseline) - Below (Month 7) | 1 | 2
  RBC, Below (baseline) - Within (Month 7): number analyzed (Participants) | 5 | 5
  RBC, Below (baseline) - Within (Month 7) | 4 | 3
  RBC, Below (baseline) - Above (Month 7): number analyzed (Participants) | 5 | 5
  RBC, Below (baseline) - Above (Month 7) | 0 | 0
  RBC, Within (baseline) - Below (Month 7): number analyzed (Participants) | 68 | 65
  RBC, Within (baseline) - Below (Month 7) | 4 | 4
  RBC, Within (baseline) - Within (Month 7): number analyzed (Participants) | 68 | 65
  RBC, Within (baseline) - Within (Month 7) | 63 | 61
  RBC, Within (baseline) - Above (Month 7): number analyzed (Participants) | 68 | 65
  RBC, Within (baseline) - Above (Month 7) | 1 | 0
  RBC, Above (baseline) - Below (Month 7): number analyzed (Participants) | 0 | 2
  RBC, Above (baseline) - Below (Month 7) |  | 0
  RBC, Above (baseline) - Within (Month 7): number analyzed (Participants) | 0 | 2
  RBC, Above (baseline) - Within (Month 7) |  | 1
  RBC, Above (baseline) - Above (Month 7): number analyzed (Participants) | 0 | 2
  RBC, Above (baseline) - Above (Month 7) |  | 1
  HCT, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 1 | 0
  HCT, Unknown (baseline) - Below (Month 7) | 0 |
  HCT, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 1 | 0
  HCT, Unknown (baseline) - Within (Month 7) | 0 |
  HCT, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 1 | 0
  HCT, Unknown (baseline) - Above (Month 7) | 1 |
  HCT, Below (baseline) - Below (Month 7): number analyzed (Participants) | 26 | 24
  HCT, Below (baseline) - Below (Month 7) | 15 | 15
  HCT, Below (baseline) - Within (Month 7): number analyzed (Participants) | 26 | 24
  HCT, Below (baseline) - Within (Month 7) | 11 | 9
  HCT, Below (baseline) - Above (Month 7): number analyzed (Participants) | 26 | 24
  HCT, Below (baseline) - Above (Month 7) | 0 | 0
  HCT, Within (baseline) - Below (Month 7): number analyzed (Participants) | 44 | 44
  HCT, Within (baseline) - Below (Month 7) | 2 | 4
  HCT, Within (baseline) - Within (Month 7): number analyzed (Participants) | 44 | 44
  HCT, Within (baseline) - Within (Month 7) | 41 | 40
  HCT, Within (baseline) - Above (Month 7): number analyzed (Participants) | 44 | 44
  HCT, Within (baseline) - Above (Month 7) | 1 | 0
  HCT, Above (baseline) - Below (Month 7): number analyzed (Participants) | 3 | 4
  HCT, Above (baseline) - Below (Month 7) | 0 | 0
  HCT, Above (baseline) - Within (Month 7): number analyzed (Participants) | 3 | 4
  HCT, Above (baseline) - Within (Month 7) | 3 | 4
  HCT, Above (baseline) - Above (Month 7): number analyzed (Participants) | 3 | 4
  HCT, Above (baseline) - Above (Month 7) | 0 | 0
  HGB, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 1 | 0
  HGB, Unknown (baseline) - Below (Month 7) | 0 |
  HGB, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 1 | 0
  HGB, Unknown (baseline) - Within (Month 7) | 0 |
  HGB, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 1 | 0
  HGB, Unknown (baseline) - Above (Month 7) | 1 |
  HGB, Below (baseline) - Below (Month 7): number analyzed (Participants) | 21 | 14
  HGB, Below (baseline) - Below (Month 7) | 10 | 7
  HGB, Below (baseline) - Within (Month 7): number analyzed (Participants) | 21 | 14
  HGB, Below (baseline) - Within (Month 7) | 11 | 7
  HGB, Below (baseline) - Above (Month 7): number analyzed (Participants) | 21 | 14
  HGB, Below (baseline) - Above (Month 7) | 0 | 0
  HGB, Within (baseline) - Below (Month 7): number analyzed (Participants) | 47 | 52
  HGB, Within (baseline) - Below (Month 7) | 1 | 7
  HGB, Within (baseline) - Within (Month 7): number analyzed (Participants) | 47 | 52
  HGB, Within (baseline) - Within (Month 7) | 40 | 44
  HGB, Within (baseline) - Above (Month 7): number analyzed (Participants) | 47 | 52
  HGB, Within (baseline) - Above (Month 7) | 6 | 1
  HGB, Above (baseline) - Below (Month 7): number analyzed (Participants) | 5 | 6
  HGB, Above (baseline) - Below (Month 7) | 0 | 0
  HGB, Above (baseline) - Within (Month 7): number analyzed (Participants) | 5 | 6
  HGB, Above (baseline) - Within (Month 7) | 3 | 5
  HGB, Above (baseline) - Above (Month 7): number analyzed (Participants) | 5 | 6
  HGB, Above (baseline) - Above (Month 7) | 2 | 1
  WBC, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 1 | 0
  WBC, Unknown (baseline) - Below (Month 7) | 0 |
  WBC, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 1 | 0
  WBC, Unknown (baseline) - Within (Month 7) | 1 |
  WBC, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 1 | 0
  WBC, Unknown (baseline) - Above (Month 7) | 0 |
  WBC, Below (baseline) - Below (Month 7): number analyzed (Participants) | 5 | 7
  WBC, Below (baseline) - Below (Month 7) | 3 | 4
  WBC, Below (baseline) - Within (Month 7): number analyzed (Participants) | 5 | 7
  WBC, Below (baseline) - Within (Month 7) | 2 | 3
  WBC, Below (baseline) - Above (Month 7): number analyzed (Participants) | 5 | 7
  WBC, Below (baseline) - Above (Month 7) | 0 | 0
  WBC, Within (baseline) - Below (Month 7): number analyzed (Participants) | 63 | 58
  WBC, Within (baseline) - Below (Month 7) | 1 | 7
  WBC, Within (baseline) - Within (Month 7): number analyzed (Participants) | 63 | 58
  WBC, Within (baseline) - Within (Month 7) | 59 | 48
  WBC, Within (baseline) - Above (Month 7): number analyzed (Participants) | 63 | 58
  WBC, Within (baseline) - Above (Month 7) | 3 | 3
  WBC, Above (baseline) - Below (Month 7): number analyzed (Participants) | 5 | 7
  WBC, Above (baseline) - Below (Month 7) | 0 | 0
  WBC, Above (baseline) - Within (Month 7): number analyzed (Participants) | 5 | 7
  WBC, Above (baseline) - Within (Month 7) | 3 | 5
  WBC, Above (baseline) - Above (Month 7): number analyzed (Participants) | 5 | 7
  WBC, Above (baseline) - Above (Month 7) | 2 | 2
  LYM, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 1 | 0
  LYM, Unknown (baseline) - Below (Month 7) | 0 |
  LYM, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 1 | 0
  LYM, Unknown (baseline) - Within (Month 7) | 1 |
  LYM, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 1 | 0
  LYM, Unknown (baseline) - Above (Month 7) | 0 |
  LYM, Below (baseline) - Below (Month 7): number analyzed (Participants) | 7 | 10
  LYM, Below (baseline) - Below (Month 7) | 5 | 6
  LYM, Below (baseline) - Within (Month 7): number analyzed (Participants) | 7 | 10
  LYM, Below (baseline) - Within (Month 7) | 1 | 3
  LYM, Below (baseline) - Above (Month 7): number analyzed (Participants) | 7 | 10
  LYM, Below (baseline) - Above (Month 7) | 1 | 1
  LYM, Within (baseline) - Below (Month 7): number analyzed (Participants) | 49 | 42
  LYM, Within (baseline) - Below (Month 7) | 6 | 5
  LYM, Within (baseline) - Within (Month 7): number analyzed (Participants) | 49 | 42
  LYM, Within (baseline) - Within (Month 7) | 37 | 36
  LYM, Within (baseline) - Above (Month 7): number analyzed (Participants) | 49 | 42
  LYM, Within (baseline) - Above (Month 7) | 6 | 1
  LYM, Above (baseline) - Below (Month 7): number analyzed (Participants) | 17 | 20
  LYM, Above (baseline) - Below (Month 7) | 1 | 1
  LYM, Above (baseline) - Within (Month 7): number analyzed (Participants) | 17 | 20
  LYM, Above (baseline) - Within (Month 7) | 10 | 8
  LYM, Above (baseline) - Above (Month 7): number analyzed (Participants) | 17 | 20
  LYM, Above (baseline) - Above (Month 7) | 6 | 11
  MONO, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 1 | 0
  MONO, Unknown (baseline) - Below (Month 7) | 1 |
  MONO, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 1 | 0
  MONO, Unknown (baseline) - Within (Month 7) | 0 |
  MONO, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 1 | 0
  MONO, Unknown (baseline) - Above (Month 7) | 0 |
  MONO, Below (baseline) - Below (Month 7): number analyzed (Participants) | 8 | 9
  MONO, Below (baseline) - Below (Month 7) | 2 | 4
  MONO, Below (baseline) - Within (Month 7): number analyzed (Participants) | 8 | 9
  MONO, Below (baseline) - Within (Month 7) | 6 | 4
  MONO, Below (baseline) - Above (Month 7): number analyzed (Participants) | 8 | 9
  MONO, Below (baseline) - Above (Month 7) | 0 | 1
  MONO, Within (baseline) - Below (Month 7): number analyzed (Participants) | 53 | 54
  MONO, Within (baseline) - Below (Month 7) | 4 | 3
  MONO, Within (baseline) - Within (Month 7): number analyzed (Participants) | 53 | 54
  MONO, Within (baseline) - Within (Month 7) | 49 | 51
  MONO, Within (baseline) - Above (Month 7): number analyzed (Participants) | 53 | 54
  MONO, Within (baseline) - Above (Month 7) | 0 | 0
  MONO, Above (baseline) - Below (Month 7): number analyzed (Participants) | 12 | 9
  MONO, Above (baseline) - Below (Month 7) | 0 | 0
  MONO, Above (baseline) - Within (Month 7): number analyzed (Participants) | 12 | 9
  MONO, Above (baseline) - Within (Month 7) | 11 | 7
  MONO, Above (baseline) - Above (Month 7): number analyzed (Participants) | 12 | 9
  MONO, Above (baseline) - Above (Month 7) | 1 | 2
  NEU, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 1 | 0
  NEU, Unknown (baseline) - Below (Month 7) | 0 |
  NEU, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 1 | 0
  NEU, Unknown (baseline) - Within (Month 7) | 1 |
  NEU, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 1 | 0
  NEU, Unknown (baseline) - Above (Month 7) | 0 |
  NEU, Below (baseline) - Below (Month 7): number analyzed (Participants) | 16 | 21
  NEU, Below (baseline) - Below (Month 7) | 5 | 10
  NEU, Below (baseline) - Within (Month 7): number analyzed (Participants) | 16 | 21
  NEU, Below (baseline) - Within (Month 7) | 10 | 10
  NEU, Below (baseline) - Above (Month 7): number analyzed (Participants) | 16 | 21
  NEU, Below (baseline) - Above (Month 7) | 1 | 1
  NEU, Within (baseline) - Below (Month 7): number analyzed (Participants) | 53 | 45
  NEU, Within (baseline) - Below (Month 7) | 4 | 4
  NEU, Within (baseline) - Within (Month 7): number analyzed (Participants) | 53 | 45
  NEU, Within (baseline) - Within (Month 7) | 43 | 35
  NEU, Within (baseline) - Above (Month 7): number analyzed (Participants) | 53 | 45
  NEU, Within (baseline) - Above (Month 7) | 6 | 6
  NEU, Above (baseline) - Below (Month 7): number analyzed (Participants) | 4 | 6
  NEU, Above (baseline) - Below (Month 7) | 0 | 1
  NEU, Above (baseline) - Within (Month 7): number analyzed (Participants) | 4 | 6
  NEU, Above (baseline) - Within (Month 7) | 2 | 2
  NEU, Above (baseline) - Above (Month 7): number analyzed (Participants) | 4 | 6
  NEU, Above (baseline) - Above (Month 7) | 2 | 3
  PLA, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 2 | 0
  PLA, Unknown (baseline) - Below (Month 7) | 0 |
  PLA, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 2 | 0
  PLA, Unknown (baseline) - Within (Month 7) | 2 |
  PLA, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 2 | 0
  PLA, Unknown (baseline) - Above (Month 7) | 0 |
  PLA, Below (baseline) - Below (Month 7): number analyzed (Participants) | 0 | 2
  PLA, Below (baseline) - Below (Month 7) |  | 0
  PLA, Below (baseline) - Within (Month 7): number analyzed (Participants) | 0 | 2
  PLA, Below (baseline) - Within (Month 7) |  | 2
  PLA, Below (baseline) - Above (Month 7): number analyzed (Participants) | 0 | 2
  PLA, Below (baseline) - Above (Month 7) |  | 0
  PLA, Within (baseline) - Below (Month 7): number analyzed (Participants) | 60 | 55
  PLA, Within (baseline) - Below (Month 7) | 0 | 0
  PLA, Within (baseline) - Within (Month 7): number analyzed (Participants) | 60 | 55
  PLA, Within (baseline) - Within (Month 7) | 56 | 53
  PLA, Within (baseline) - Above (Month 7): number analyzed (Participants) | 60 | 55
  PLA, Within (baseline) - Above (Month 7) | 4 | 2
  PLA, Above (baseline) - Below (Month 7): number analyzed (Participants) | 12 | 15
  PLA, Above (baseline) - Below (Month 7) | 0 | 0
  PLA, Above (baseline) - Within (Month 7): number analyzed (Participants) | 12 | 15
  PLA, Above (baseline) - Within (Month 7) | 7 | 8
  PLA, Above (baseline) - Above (Month 7): number analyzed (Participants) | 12 | 15
  PLA, Above (baseline) - Above (Month 7) | 5 | 7
  BUN, Unknown (baseline) - Below (Month 7): number analyzed (Participants) | 2 | 1
  BUN, Unknown (baseline) - Below (Month 7) | 0 | 0
  BUN, Unknown (baseline) - Within (Month 7): number analyzed (Participants) | 2 | 1
  BUN, Unknown (baseline) - Within (Month 7) | 2 | 1
  BUN, Unknown (baseline) - Above (Month 7): number analyzed (Participants) | 2 | 1
  BUN, Unknown (baseline) - Above (Month 7) | 0 | 0
  BUN, Below (baseline) - Below (Month 7): number analyzed (Participants) | 12 | 4
  BUN, Below (baseline) - Below (Month 7) | 5 | 0
  BUN, Below (baseline) - Within (Month 7): number analyzed (Participants) | 12 | 4
  BUN, Below (baseline) - Within (Month 7) | 7 | 4
  BUN, Below (baseline) - Above (Month 7): number analyzed (Participants) | 12 | 4
  BUN, Below (baseline) - Above (Month 7) | 0 | 0
  BUN, Within (baseline) - Below (Month 7): number analyzed (Participants) | 52 | 61
  BUN, Within (baseline) - Below (Month 7) | 4 | 10
  BUN, Within (baseline) - Within (Month 7): number analyzed (Participants) | 52 | 61
  BUN, Within (baseline) - Within (Month 7) | 47 | 51
  BUN, Within (baseline) - Above (Month 7): number analyzed (Participants) | 52 | 61
  BUN, Within (baseline) - Above (Month 7) | 1 | 0
  BUN, Above (baseline) - Below (Month 7): number analyzed (Participants) | 6 | 6
  BUN, Above (baseline) - Below (Month 7) | 0 | 0
  BUN, Above (baseline) - Within (Month 7): number analyzed (Participants) | 6 | 6
  BUN, Above (baseline) - Within (Month 7) | 6 | 6
  BUN, Above (baseline) - Above (Month 7): number analyzed (Participants) | 6 | 6
  BUN, Above (baseline) - Above (Month 7) | 0 | 0

7. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs) From Day 0 up to Month 7
Description: SAEs assessed included medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 up to Month 7 (i.e. from first vaccination at Day 0 up to 30 days after the second vaccination at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants | 0 | 2

8. Primary Outcome: Number of Subjects With AEs and SAEs Leading to Withdrawal From Day 0 up to Month 7
Description: The number of subjects with AEs and SAEs leading to premature discontinuation of the study was assessed.
Time Frame: From Day 0 up to Month 7 (i.e. from first vaccination at Day 0 up to 30 days after the second vaccination at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants | 0 | 0

9. Primary Outcome: Number of Subjects With Potential Immune-mediated Diseases (pIMDs) From Day 0 up to Month 7
Description: pIMDs were defined as a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which might or might not have an autoimmune aetiology.
Time Frame: From Day 0 up to Month 7 (i.e. from first vaccination at Day 0 up to 30 days after the second vaccination at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants | 0 | 0

10. Primary Outcome: Number of Subjects With Medically Significant Conditions (MSCs) From Day 0 up to Month 7
Description: MSCs were defined as AEs prompting emergency room or physician visits that were not related to common diseases or were not routine visits for physical examination or vaccination and as SAEs that were not related to common diseases. Common diseases included: upper respiratory tract infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections and injury.
Time Frame: From Day 0 up to Month 7 (i.e. from first vaccination at Day 0 up to 30 days after the second vaccination at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants | 37 | 28

11. Primary Outcome: Number of Seroconverted Subjects for HPV-16 and HPV-18 Antigens at Month 7
Description: Seroconversion was defined as a titer greater than or equal to the cut-off value in the serum of seronegative subjects, defined as subjects who had an antibody titer below the cut-off value before vaccination. Titers were measured by Enzyme Linked Immunosorbent Assay (ELISA) and the cut-offs were 19 ELISA Units per milliliter (EU/mL) for HPV-16 and 18 EU/mL for HPV-18.
Time Frame: At Month 7 (i.e. 30 days after the vaccination at Month 6)
Population: The analysis was performed on the According-to-protocol (ATP) cohort for immunogenicity at Month 7, which included all eligible subjects (i.e. meeting all eligibility criteria, complying with the procedures defined in the protocol) for whom data concerning immunogenicity outcome measures were available at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 64 | 44
Participants
  Anti-HPV-16: number analyzed (Participants) | 64 | 43
  Anti-HPV-16 | 64 | 1
  Anti-HPV-18: number analyzed (Participants) | 62 | 44
  Anti-HPV-18 | 62 | 1

12. Primary Outcome: Anti-HPV-16/18 Antibody Concentrations at Month 7
Description: Antibody concentrations were assessed by ELISA and expressed as geometric mean concentrations (GMCs) in EU/mL.
Time Frame: At Month 7 (i.e. 30 days after the vaccination at Month 6)
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 64 | 44
EU/mL
  Anti-HPV-16: number analyzed (Participants) | 64 | 43
  Anti-HPV-16 | 20080.0 [16831.8 to 23954.9] | 10.4 [8.7 to 12.5]
  Anti-HPV-18: number analyzed (Participants) | 62 | 44
  Anti-HPV-18 | 10621.8 [8865.3 to 12726.3] | 9.6 [8.4 to 11.1]

13. Secondary Outcome: Number of Seroconverted Subjects for HPV-16 and HPV-18 Antigens at Month 7, Month 12 (for Both Groups) and at Month 18, Month 24 and Month 36 (Only for Cervarix Group)
Description: Seroconversion was defined as a titer greater than or equal to the cut-off value in the serum of seronegative subjects, defined as subjects who had an antibody titer below the cut-off value before vaccination. Titers were measured by ELISA and the cut-offs were 19 EU/mL for HPV-16 and 18 EU/mL for HPV-18. Note: Month 7 data are also reported in the Primary outcome measure.
Time Frame: At Month 7, Month 12 (for both groups) and at Month 18, Month 24 and Month 36 (only for Cervarix Group)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all eligible subjects for whom data concerning immunogenicity outcome measures were available at the specified time point. Priorix+Infanrix Group data were only tabulated for the time points up to Month 12, since the follow-up phase for this group ended at Month 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 67 | 49
Participants
  Anti-HPV-16, Month 7: number analyzed (Participants) | 64 | 43
  Anti-HPV-16, Month 7 | 64 | 1
  Anti-HPV-16, Month 12: number analyzed (Participants) | 65 | 48
  Anti-HPV-16, Month 12 | 65 | 1
  Anti-HPV-16, Month 18: number analyzed (Participants) | 66 | 0
  Anti-HPV-16, Month 18 | 66 |
  Anti-HPV-16, Month 24: number analyzed (Participants) | 67 | 0
  Anti-HPV-16, Month 24 | 67 |
  Anti-HPV-16, Month 36: number analyzed (Participants) | 67 | 0
  Anti-HPV-16, Month 36 | 67 |
  Anti-HPV-18, Month 7: number analyzed (Participants) | 62 | 44
  Anti-HPV-18, Month 7 | 62 | 1
  Anti-HPV-18, Month 12: number analyzed (Participants) | 63 | 49
  Anti-HPV-18, Month 12 | 63 | 0
  Anti-HPV-18, Month 18: number analyzed (Participants) | 64 | 0
  Anti-HPV-18, Month 18 | 64 |
  Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 0
  Anti-HPV-18, Month 24 | 65 |
  Anti-HPV-18, Month 36: number analyzed (Participants) | 65 | 0
  Anti-HPV-18, Month 36 | 65 |

14. Secondary Outcome: Anti-HPV-16 and Anti-HPV-18 Antibody Concentrations at Month 7, Month 12 (for Both Groups) and at Month 18, Month 24 and Month 36 (Only for Cervarix Group)
Description: Antibody concentrations were assessed by ELISA and expressed as GMCs in EU/mL. Note: Month 7 data are also reported in the Primary outcome measure.
Time Frame: At Month 7, Month 12 (for both groups) and at Month 18, Month 24 and Month 36 (only for Cervarix Group)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 67 | 49
EU/mL
  Anti-HPV-16, Month 7: number analyzed (Participants) | 64 | 43
  Anti-HPV-16, Month 7 | 20080.0 [16831.8 to 23954.9] | 10.4 [8.7 to 12.5]
  Anti-HPV-16, Month 12: number analyzed (Participants) | 65 | 48
  Anti-HPV-16, Month 12 | 3246.5 [2617.4 to 4026.8] | 9.7 [9.3 to 10.2]
  Anti-HPV-16, Month 18: number analyzed (Participants) | 66 | 0
  Anti-HPV-16, Month 18 | 2800.5 [2325.8 to 3372.0] |
  Anti-HPV-16, Month 24: number analyzed (Participants) | 67 | 0
  Anti-HPV-16, Month 24 | 1951.9 [1553.7 to 2452.2] |
  Anti-HPV-16, Month 36: number analyzed (Participants) | 67 | 0
  Anti-HPV-16, Month 36 | 1680.6 [1384.2 to 2040.4] |
  Anti-HPV-18, Month 7: number analyzed (Participants) | 62 | 44
  Anti-HPV-18, Month 7 | 10621.8 [8865.3 to 12726.3] | 9.6 [8.4 to 11.1]
  Anti-HPV-18, Month 12: number analyzed (Participants) | 63 | 49
  Anti-HPV-18, Month 12 | 1216.6 [953.1 to 1553.0] | 9.0 [9.0 to 9.0]
  Anti-HPV-18, Month 18: number analyzed (Participants) | 64 | 0
  Anti-HPV-18, Month 18 | 802.9 [632.4 to 1019.5] |
  Anti-HPV-18, Month 24: number analyzed (Participants) | 65 | 0
  Anti-HPV-18, Month 24 | 766.6 [603.3 to 974.2] |
  Anti-HPV-18, Month 36: number analyzed (Participants) | 65 | 0
  Anti-HPV-18, Month 36 | 536.4 [420.6 to 684.0] |

15. Secondary Outcome: Number of Seropositive Subjects for Measles Antigen
Description: A seropositive subject was defined as a subject whose anti-measles antibody titer was equal to or above (≥) 150 milli-International Units per milliliter (mIU/mL), as assessed by ELISA.
Time Frame: At Day 0 and Day 42 (i.e. 42 days after the vaccination at Day 0)
Population: The analysis was performed on the ATP cohort for immunogenicity at Day 42, which included all eligible subjects (i.e. meeting all eligibility criteria, complying with the procedures defined in the protocol) for whom data concerning immunogenicity outcome measures were available at Day 42.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 68 | 58
Participants
  Anti-measles, Day 0: number analyzed (Participants) | 66 | 55
  Anti-measles, Day 0 | 65 | 50
  Anti-measles, Day 42 | 67 | 58

16. Secondary Outcome: Anti-measles Antibody Concentrations
Description: Anti-measles antibody concentrations were measured by ELISA, expressed as GMCs, in mIU/mL. The cut-off of the assay was an anti-measles antibody concentration ≥ 150 mIU/mL.
Time Frame: At Day 0 and Day 42 (i.e. 42 days after the vaccination at Day 0)
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 68 | 58
mIU/mL
  Anti-measles, Day 0: number analyzed (Participants) | 66 | 55
  Anti-measles, Day 0 | 1029.8 [852.8 to 1243.6] | 694.8 [524.0 to 921.3]
  Anti-measles, Day 42 | 897.1 [748.8 to 1074.8] | 2512.3 [2140.3 to 2949.0]

17. Secondary Outcome: Number of Seropositive Subjects for Mumps Antigen
Description: A seropositive subject was defined as a subject whose anti-mumps antibody titer was equal to or above (≥) 231 U/mL, as assessed by ELISA.
Time Frame: At Day 0 and Day 42 (i.e. 42 days after the vaccination at Day 0)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 68 | 58
Participants
  Anti-mumps, Day 0: number analyzed (Participants) | 66 | 55
  Anti-mumps, Day 0 | 64 | 50
  Anti-mumps, Day 42 | 66 | 57

18. Secondary Outcome: Anti-mumps Antibody Concentrations
Description: Anti-mumps antibody concentrations were measured by ELISA, expressed as GMCs, in U/mL. The cut-off of the assay was an anti-mumps antibody concentration ≥ 231 U/mL.
Time Frame: At Day 0 and Day 42 (i.e. 42 days after the vaccination at Day 0)
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 68 | 58
U/mL
  Anti-mumps, Day 0: number analyzed (Participants) | 66 | 55
  Anti-mumps, Day 0 | 3613.7 [2742.1 to 4762.4] | 2142.6 [1492.7 to 3075.5]
  Anti-mumps, Day 42 | 3594.1 [2749.1 to 4698.8] | 7001.1 [5414.9 to 9052.1]

19. Secondary Outcome: Number of Seropositive Subjects for Rubella Antigen
Description: A seropositive subject was defined as a subject whose anti-rubella antibody titer was ≥ 4 IU/mL, as assessed by ELISA.
Time Frame: At Day 0 and Day 42 (i.e. 42 days after the vaccination at Day 0)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 68 | 58
Participants
  Anti-rubella, Day 0: number analyzed (Participants) | 66 | 55
  Anti-rubella, Day 0 | 66 | 53
  Anti-rubella, Day 42 | 68 | 58

20. Secondary Outcome: Anti-rubella Antibody Concentrations
Description: Anti-rubella antibody concentrations were measured by ELISA, expressed as GMCs, in IU/mL. The cut-off of the assay was an anti-rubella antibody concentration ≥ 4 IU/mL.
Time Frame: At Day 0 and Day 42 (i.e. 42 days after the vaccination at Day 0)
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 68 | 58
IU/mL
  Anti-rubella, Day 0: number analyzed (Participants) | 66 | 55
  Anti-rubella, Day 0 | 82.0 [69.4 to 96.8] | 48.9 [36.3 to 65.9]
  Anti-rubella, Day 42 | 79.3 [67.3 to 93.6] | 124.2 [107.0 to 144.2]

21. Secondary Outcome: Number of Seroprotected Subjects Against Diphtheria and Tetanus Antigens
Description: A seroprotected subject against diphtheria antigen was defined as a subject with an anti-diphtheria (anti-D) antibody concentration ≥ the cut-off of 0.1 IU/mL, as measured by ELISA.
  A seroprotected subject against tetanus antigen was defined as a subject with an anti-tetanus (anti-T) antibody concentration ≥ the cut-off of 0.1 IU/mL, as measured by ELISA.
Time Frame: At Month 7 (i.e. 30 days after the vaccination at Month 6)
Population: The analysis was performed on the ATP cohort for immunogenicity at Month 7, which included all eligible subjects (i.e. meeting all eligibility criteria, complying with the procedures defined in the protocol) for whom data concerning immunogenicity outcome measures were available at Month 7.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 65 | 47
Participants
  Anti-D | 45 | 47
  Anti-T | 60 | 47

22. Secondary Outcome: Number of Subjects With pIMDs From Day 0 up to Month 12
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which might or might not have an autoimmune aetiology.
Time Frame: From Day 0 up to Month 12 (i.e. from first vaccination at Day 0 up to 6 months after the second vaccination at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants | 0 | 0

23. Secondary Outcome: Number of Subjects With MSCs From Day 0 up to Month 12
Description: as for outcome 10
Time Frame: From Day 0 up to Month 12 (i.e. from first vaccination at Day 0 up to 6 months after the second vaccination at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants | 38 | 29

24. Secondary Outcome: Number of Subjects With SAEs From Day 0 up to Month 12
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 up to Month 12 (i.e. from first vaccination at Day 0 up to 6 months after the second vaccination at Month 6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants | 1 | 2

25. Secondary Outcome: Number of Subjects With SAEs Related to the Investigational Products or Any Fatal SAE
Description: SAEs assessed included medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the study period (i.e. from Day 0 up to Month 12 for Priorix + Infanrix Group and from Day 0 up to Month 36 for Cervarix Group)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants
  Related SAE(s) | 0 | 0
  Fatal SAE(s) | 0 | 0

26. Secondary Outcome: Number of Subjects With AEs/SAEs Leading to Withdrawal Throughout the Study Period
Description: The number of subjects with AEs and SAEs leading to premature discontinuation of study was assessed.
Time Frame: Throughout the study period (i.e from Day 0 up to Month 12 for Priorix + Infanrix Group and from Day 0 up to Month 36 for Cervarix Group)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants | 0 | 0

27. Secondary Outcome: Number of Subjects Reporting the Intake of Concomitant Medication During the 43-day Period Following the Vaccination at Day 0
Description: Concomitant medication taken at least once during the 43-day period (i.e. from the day of vaccination up to 42 subsequent days) following the vaccination at Day 0 included: any type of medicines, antipyretics, prophylactic antipyretics and antibiotics.
Time Frame: During the 43-day period (i.e. from the day of vaccination up to 42 subsequent days) following the vaccination at Day 0
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants
  Any medication | 45 | 36
  Any antipyretic | 29 | 24
  Prophylactic antipyretic | 0 | 0
  Any antibiotic | 18 | 10

28. Secondary Outcome: Number of Subjects Reporting the Intake of Concomitant Medication During the 30-day Period Following the Vaccination at Month 6
Description: Concomitant medication taken at least once during the 30-day period (i.e. from the day of vaccination up to 29 subsequent days) following the vaccination at Month 6 included: any type of medicines, antipyretics, prophylactic antipyretics and antibiotics.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 71
Participants
  Any medication | 19 | 23
  Any antipyretic | 10 | 8
  Prophylactic antipyretic | 0 | 0
  Any antibiotic | 6 | 6

29. Secondary Outcome: Percentage of Subjects Completing the Vaccination Schedule in Both Groups
Description: The percentage of subjects who received the specified total number of doses (dose 1, dose 2, any dose) is reported.
Time Frame: From Day 0 up to Month 6 (i.e. from first vaccination at Day 0 up to the second vaccination at Month 6)
Population: as for outcome 3
Measure: Number; unit: Percentage of subjects
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Percentage of subjects
  Subjects receiving only 1 dose | 0 | 4.1
  Subjects receiving 2 doses | 100 | 95.9
  Subjects receiving at least 1 dose | 100 | 100

30. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related to Vaccination Solicited Fever, Measles/Rubella-like Rash, Parotid Gland Swelling and Signs of Meningism Including Febrile Convulsion
Description: Measles/Rubella-like rash: presence of macules, discoloured small patches or spots of the skin, neither elevated nor depressed below the skin's surface and/or papules, raised bumps on the skin usually below (<) 1 cm in diameter.
  Parotid/salivary gland swelling: swelling/tenderness in the mandibular/submandibular region.
  Suspected signs of meningism including febrile convulsions: febrile convulsions or any other neurological signs or symptoms indicative of meningism.
  Any = occurrence of any solicited symptom regardless of their intensity grade or relationship to vaccination. Any fever = axillary temperature equal to or above (≥) 37.5°C. Grade 3 AE = AE which prevented normal, everyday activities. Grade 3 measles/rubella-like rash = more than 150 lesions. Grade 3 parotid gland swelling = swelling with accompanying general symptoms. Grade 3 fever = axillary temperature above (>) 39.0°C. Related = any symptom assessed by the investigator as causally related to the vaccination.
Time Frame: During the 43-day period (i.e. from the day of vaccination up to 42 subsequent days) following the vaccination at Day 0
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Priorix + Infanrix Group
Number analyzed (Participants) | 74 | 74
Participants
  Any Fever | 30 | 27
  Grade 3 Fever | 7 | 2
  Related Fever | 6 | 7
  Any Measles/Rubella-like rash | 1 | 1
  Grade 3 Measles/Rubella-like rash | 0 | 0
  Related Measles/Rubella-like rash | 1 | 1
  Any Parotid gland swelling | 0 | 0
  Grade 3 Parotid gland swelling | 0 | 0
  Related Parotid gland swelling | 0 | 0
  Any Signs of meningism | 0 | 1
  Grade 3 Signs of meningism | 0 | 0
  Related Signs of meningism | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited AEs: During the 7-day period after each vaccination. Unsolicited AEs: During the 43-day period after the vaccination at Day 0 and during the 30-day period after the vaccination at Month 6. SAEs: From Day 0 up to Month 12.
Arm/Group | Cervarix Group | Priorix + Infanrix Group
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/74
Serious Adverse Events (participants affected / at risk) | 1/74 | 2/74
Other Adverse Events (participants affected / at risk) | 70/74 | 65/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix Group (N=74) | Priorix + Infanrix Group (N=74)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cervarix Group (N=74) | Priorix + Infanrix Group (N=74)
Pain (General disorders) | 54 (88) | 40 (51)
Swelling (General disorders) | 19 (22) | 18 (21)
Fatigue (General disorders) | 15 (17) | 10 (14)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acarodermatitis (Infections and infestations) | 2 (2) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (15) | 11 (16)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 21 (24) | 13 (15)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 18 (22) | 18 (19)
Eye allergy (Eye disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 7 (7)
Gastrointestinal disorder (Gastrointestinal disorders) | 11 (11) | 16 (21)
Giardiasis (Infections and infestations) | 1 (1) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 18 (25) | 25 (35)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 3 (3) | 0 (0)
Infection parasitic (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 22 (31) | 19 (24)
Lice infestation (Infections and infestations) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Meningism (Nervous system disorders) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 21 (26) | 14 (20)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 24 (28) | 27 (33)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 6 (6) | 4 (4)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 36 (39) | 33 (39)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 16 (23) | 15 (16)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 10 (10) | 7 (7)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vulvovaginitis (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.